## **Notification of Approval**

Date: 3 July 2025

Study ID: Pro00153815

Principal Investigator: Lisa Hartling

Study Title: Language translation of knowledge mobilization resources: A randomized trial

Approval Expiry Date: Thursday, July 2, 2026

Sponsor/Funding Agency:

Alberta Innovates Health Solutions

AIHS

Canada

Thank you for submitting the above study to the Research Ethics Board 2. Your application has been reviewed and approved on behalf of the committee.

## **Approved Documents:**

#### Recruitment Materials

RecruitmentBlurb 27JUN2025 V1.docx

RecruitmentPoster 27JUN2025 V1.pdf

EmailScript\_Stakeholders\_27JUN2025\_V1.docx

### Letter of Initial Contact

LetterofInitialContact 27JUN2025 V1.docx

#### **Consent Forms**

StudyInformationLetter\_27JUN2025\_V1.docx

# Questionnaires, Cover Letters, Surveys, Tests, Interview Scripts, etc.

REDCapSurveyTemplate\_27JUN2025\_V1.docx

### Protocol/Research Proposal

Al\_StudyProtocol\_27JUN2025 V1.docx

#### Other Documents

GiftCardLog 27JUN2025.xlsx

GiftCardMessage 27JUN2025 V1.docx

Translated KM Resources.pdf

Any proposed changes to the study must be submitted to the REB for approval prior to implementation. A renewal report must be submitted next year prior to the expiry of this approval if your study still requires ethics approval. If you do not renew on or before the renewal expiry date, you will have to re-submit an ethics

application.

Approval by the REB does not constitute authorization to initiate the conduct of this research. The Principal Investigator is responsible for ensuring required approvals from other involved organizations (e.g., local universities/colleges, community organizations, school boards) are obtained, before the research begins.

Sincerely,

Ubaka Ogbogu, LLB, BL, LLM, SJD Chair, Research Ethics Board 2

Note: This correspondence includes an electronic signature (validation and approval via an online system).